CLINICAL TRIAL: NCT03154372
Title: Deliberate Practice With Validated Metrics Improves Skill Acquisition in Performance of Ultrasound Guided Peripheral Nerve Block in a Simulated Setting
Brief Title: Deliberate Practice With Validated Metrics Improves Skills Acquisition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Osman Ahmed, Principal Investigator, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 27th April, 2016.
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Educational Problems

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- deliberate practice (Other): expert supervised practice with validated metrics
  Interventions: Other: Expert supervised practice with validated metrics
- self-guided practice (Other): self guided practice with validated metrics
  Interventions: Other: self guided practice with validated metrics

INTERVENTIONS:
Other: Expert supervised practice with validated metrics
  Arms: deliberate practice
Other: self guided practice with validated metrics
  Arms: self-guided practice

SUMMARY:
Purpose:

The aim of this study was to compare the effects of deliberate vs. self-guided practices on acquiring needling skills by novice learners.

Methods:

Eighteen medical students were randomized to deliberate or self-guided practices groups. Following a learning phase, subjects attempted to perform a predefined task, which entitled advancing a needle towards a target on a phantom gel under ultrasound guidance. Subsequently, all subjects practiced performing the task using previously validated metrics. Subjects in the deliberate practice group were coached by an expert anesthesiologist and practiced each metric until it was satisfactorily performed based on the supervising anesthesiologist assessment. Immediately after completing the practice, all subjects attempted to perform same task, and on the following day, made two further attempts in succession. Two trained consultant anesthesiologists will use the metrics to independently score the video-recorded performances.

DETAILED DESCRIPTION:
Safe performance of ultrasound-guided peripheral nerve blocks (PNB) requires competence across a range of technical and nontechnical skills. Correct placement of a needle close to a nerve or plexus is critical to safe and successful procedure performance. Failure to maintain needle visibility while in forward motion may cause iatrogenic injury to nerves and surrounding structures, and is a "quality compromising" behavior in the early part of novice learning curve. Skills related to needle guidance are difficult to learn, as they require integration of multiple cognitive and psychomotor elements.

The objective of this study was to compare the effects of expert supervised deliberate practice with validated metrics vs. self-guided practice on novice needling skill acquisition as evaluated by the number of steps completed and errors made.

Methods

Having obtained informed written consent from each, eighteen 3rd and 4th year medical students with no previous experience of ultrasound-guided procedures were recruited. Each student provided demographic information on his or her age, gender and handedness. All subjects will attend a didactic lecture (learning phase) delivered in standard fashion by one investigator. This included outlines of ultrasound physics, scanning and practical techniques.

Subsequently, subjects will be randomly allocated using computer generated random numbers to one of two groups; self-guided practice (SP) and deliberate practice (DP). Approximately 24 hours after completion of the learning phase each subject will attempt to perform the following set of tasks (baseline assessment).

Task description (i) Perform ultrasonography of the phantom provided to identify embedded objects.

(ii) Identify verbally the structure at the 8 O'clock position (in reference to the ultrasound training block model) and surrounding structures.

(iii) Once the ultrasound image is deemed optimal, advance a 50 mm, 20 gauge block needle provided under ultrasound guidance towards the object at the 8 O'clock position.

(iv) Once the needle tip is deemed close enough to the object, inject 0.5 ml of saline.

Following the first set of tasks (baseline assessment), all subjects were allowed to practice the task using the list of metrics and according to their random group allocation.

Methods of practice allowed SP Group: An investigator will provide subjects in this group a list of metrics (steps and errors) extracted from a previously validated tool. They will be allowed to practice the task using the metrics list. When the subject declares readiness to progress to the assessment, training will be complete.

DP Group: A trained consultant anesthesiologist (expert in ultrasound-guided PNB and who regularly undertakes training of novices in these procedures) will supervise deliberate practice to each subject in this group using the metrics list. Subjects in this group will practice each item of the metric list until it is satisfactorily performed as assessed by the supervising anesthesiologist at which time training is deemed complete.

Immediately after completion of either self-guided practice or deliberate practice (training phase), all subjects in both groups will attempt the same task above (assessment 1). All subjects will also attempt the same task twice in succession on the following day (assessment 2 and 3).

All performances (baseline and 1- 3) will be videotaped using a head-mounted camera placed on subject's head. The first person video and ultrasound images record concurrently (time synchronized).

Two consultant anesthesiologists (each expert in performing PNB and who regularly train novices) will independently score the videos using the composite metrics list for number of steps completed and number of errors made (primary outcome).

Data and Statistical Analysis Differences in performances between the two groups for both primary and secondary outcomes will be examined for significance with one-factor analyses of variance (ANOVA).

The inter rater reliability (IRR) will be calculated according to proportionate agreement between the two video assessors "number of agreements/number of [agreements+disagreements]". IRR is considered to be acceptable if it was ≥ 0.8. Scores from both video assessors will be averaged to calculate the number of steps completed and number of errors made (primary outcome).

ELIGIBILITY:
Inclusion Criteria:

* 3rd and 4th year medical students

Exclusion Criteria:

* previous performance of ultrasound guided procedures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
number of steps completed and errors made | up to 24 hours
  averaged score of the two video assessors is calculated for number of steps completed and error made